CLINICAL TRIAL: NCT00818558
Title: Evaluation of the Value Forecasts of the Identification of the Circulating Tumoral Cells (CTC) in the Broncho-lung Carcinomas Not in Small Cells of Stages I and II by the Method ISET (Insulation by Size of Epithelial Tumor Cells)
Brief Title: The Method ISET (Insulation by Size of Epithelial Tumor Cells)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-APN-08
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (6):
- 1 (Experimental): stade IA [pT1 N0M0]
  Interventions: Biological: ISET Methode
- 2 (Experimental): stade IB [pT2 N0M0]
  Interventions: Biological: ISET Methode
- 3 (Experimental): stade IIA [pTI N1M0]
  Interventions: Biological: ISET Methode
- 4 (Experimental): stade IIB [pT2 N1 et T3N0M0]
  Interventions: Biological: ISET Methode
- 5 (Experimental): control groupe [tabagic subject]
  Interventions: Biological: ISET Methode
- 6 (Experimental): Control group B [intervention for a pulmonaire non tumoral pulmonary lesion]
  Interventions: Biological: ISET Methode

INTERVENTIONS:
Biological: ISET Methode — Sampling of blood - ISET Methode

SUMMARY:
The aim of this study is, i) to assess the presence and the frequency of CTC in NSCLC patients undergoing surgery by using cytopathological analysis after their isolation by size (ISET method), and, ii) to correlate the presence of CNHC with pTNM stage, histological subtype, and percentage of tumor cells present into the primary tumors.

DETAILED DESCRIPTION:
Lung cancer is the most prevalent neoplasm and the major cause of tumor-related mortality worldwide. Despite recent advances in the management of resected lung cancers (i.e., the use of adjuvant therapy) and more effective treatments of metastatic tumors (i.e., molecular targeted agents), the cure rate of patients with lung cancer remains low (. Histological classification of lung tumors distinguishes small (SCLC) and non-small cell lung cancers (NSCLC). Most NSCLC display three histological subtypes: adenocarcinoma, squamous cell carcinoma and large cell carcinoma. The prognosis of these three NSCLC subtypes is quite similar. In this regard, development and validation of new prognostic/predictive biomarkers from tumor tissues and biological fluids is one of the more promising domain in translational cancer research. However, the clinical impact of new biomarkers has to be carefully validated, including for NSCLC. While pTNM staging is currently the only validated prognostic factor used in NSCLC patients follow up and treatment, 25% to 50% of patients with early-stage I NSCLC show tumor recurrence following extensive tumor resection, indicating the urgent need of more sensitive prognostic markers. Furthermore, it has been reported that the presence of occult metastatic disease correlates with disease recurrence in stage I NSCLC patients. There is now a sizable body of evidence that metastases could develop from circulating tumor cells (CTC) spread in blood before or during surgery . Thus, sensitive and specific detection of CTC in blood is considered as a potentially relevant predictive biomarker for patients with NSCLC. Indeed, the main goal for preoperative detection of CTC is to identify patients with high risk of recurrence after surgery, in order to perform more adapted therapeutic strategy. Despite several studies reported about CTC detection, methodological aspects concerning sensitivity, specificity and reproducibility have prevented a clear appraisal of their clinical impact. While RT-PCR and immune-mediated methods can be very sensitive, specificity remains a critical issue for these approaches as no transcript or antigen is known at present specifically recognizing tumor cells from solid tumors . In this setting, cytopathological analysis of circulating non hematological cells (CNHC), of epithelial (CEC) and endothelial (CEN-C) origin, isolated according to their size (ISET, Isolation by Size of Epithelial Tumor cells) is considered a promising approach, as CNHC enrichment is very sensitive and cell morphology is not damaged allowing to apply classical cytopathological criteria to identify tumor cells. In this regard, ISET technology has been previously reported to allow identification of CTC in patients with liver and breast tumors. However, ISET method has never been used to detect CTC in patients with NSCLC. The aim of this study is to determine the diagnostic potential of ISET method for preoperative detection of CTC in NSCLC patients. For this purpose cytomorphological criteria have been established by a group of 10 cytologists to classify CNHC in 3 groups : i) CNHC with malignant features (CNHC-MF) , ii) CNHC with uncertain features (CNHC-UMF), and, iii) CNHC with benign features (CNHC-BF). The presence and number of these circulating cells are then correlated with pTNM, histological subtype, and percentage of tumor cells into the primary tumors.

ELIGIBILITY:
Inclusion Criteria:

For the patients:

* patient having been operated for a strong suspicion or a suspicion of a malignant tumoral hurt corresponding to a primitive carcinoma not in small cell of the lung

For the control subjects:

* Tabagical patients (between 10 and 30 packages years)
* unhurt of any malignant or mild tumoral pathology or patients that must benefit from a surgical operation for an extract of a hurt lung parenchymateuse for a not tumoral hurt

Exclusion Criteria:

* Patient with histories of cancer or the other synchronous cancer
* Patient with carcinomas with small cells, bronchiolo-alveolar carcinomas, the other types of tumors (lymphomes, sarcomas, etc.).
* Patient with neoadditives treatments
* Patient according to treatments additives others than protocols codified (in particular, platinum navelbine or gemcitabine platinum) for stages II

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of circulating tumoral Cells(Units) according to: 1) The pTNM stage 2) the histological type | immediately

SECONDARY OUTCOMES:
Specific survival and global survival, recurrence and metastasis | in 2 years, 3 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pr Hofman, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Pr Paul HOFMAN, Nice, France